CLINICAL TRIAL: NCT00926978
Title: Comparison of I-124 and I-131 Radiopharmacokinetics in Patients Who Have Well-differentiated Thyroid Cancer and Are Prepared With Recombinant Human TSH Injection (rhTSH)
Brief Title: Comparison of Iodine-124 (I-124) and Iodine-131 (I-131) Radiopharmacokinetics in Patients Prepared With Recombinant Human TSH Injection (rhTSH)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional RDRC dissolved
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Douglas Van Nostrand, Director, Nuclear Medicine Research, Medstar Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008-292
Record Dates: First submitted 2009-06-17; First posted 2009-06-24 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid; I-124
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiopharmacokinetics (Other): 1-2 mCi I-124 orally, once per day, twice total 0.9mg rhTSH intravenous injection, once per day, four total
  After TSH stimulation with Recombinant human TSH (rhTSH) for 2 days, a dose of radioactive iodine 124 ( I-124) 1.7 mCi is administrated orally and PET imaging is done for 5 continuous days including the day of the dose administration. On each day, just before imaging, 5 ml of blood is drawn.
  Patients will be randomized to either the sequence above (e.g. I-131 followed by I-124) or to the reverse sequence in which the I-124 is given first followed by the I-131. If I-124 is administered first and as long as the whole body retention is < 2% by the start of the second rhTSH stimulation, the I-124 will not interfere with the I-131.
  Interventions: Radiation: Radioactive Iodine 124

INTERVENTIONS:
Radiation: Radioactive Iodine 124 — After TSH stimulation with Recombinant human TSH (rhTSH) for 2 days, a dose of radioactive iodine 124 ( I-124) 1.7 mCi is administrated orally and PET imaging is done for 5 continuous days including the day of the dose administration. On each day, just before imaging, 5 ml of blood is drawn.
  Patients will be randomized to either the sequence above (e.g. I-131 followed by I-124) or to the reverse sequence in which the I-124 is given first followed by the I-131. If I-124 is administered first and as long as the whole body retention is < 2% by the start of the second rhTSH stimulation, the I-124 will not interfere with the I-131.
  Other Names: Sodium [124I] iodide solution in 0.02 N aqueous NaOH

SUMMARY:
This research study is to compare the radiopharmacokinetics of I-124 to the radiopharmacokinetics of I-131 in patients who have well-differentiated thyroid cancer after recombinant human thyroid-stimulating hormone (rhTSH) injection. I-131 is routinely used for imaging and dosimetry for patients with well-differentiated thyroid cancer. In this study, I-124 is administered orally in capsular form, and the radiopharmacokinetics of I-124 is compared with I-131. I-124 is another isotope of iodine, which is cyclotron-produced. I-124 has multiple advantages:

* Ideal Half-Life (4.2 days) for delayed imaging.
* High resolution tomographic imaging.
* Feasibility of quantitating lesion uptake.
* Potential of dosimetry for the planning of radioiodine therapy.

Voluntary patients will have I-124 dosimetry performed in addition to the I-131 dosimetry, which is planned as part of routine clinical care. I-124 dosimetry is composed of four parts: (1) two extra doses of injections of rhTSH, (2) the administration of I-124, (3) PET imaging, and (4) drawing blood samples.

Patients will receive two additional injections of rhTSH. This is similar to the procedure for I-131 dosimetry. Second, they will receive I-124. I-124 is similar to I-131 except I-124 decays in a different way to emit a positron so that the PET scanner can be used for imaging. I-124 is given in the form of one or several capsules, which are taken by mouth. This is also similar to I-131. Third, PET/CT imaging is done for approximately 30 minutes to one hour on five consecutive days. Radiation from PET/CT scan is far less than what they receive from a diagnostic CT scan. For the fourth part, a technologist will draw about 5 cc from the forearm on each of the five consecutive days. This is also similar to I-131.

Initially, all patients will be randomized to one of two study groups. The first group will have the I-131 dosimetry performed first followed by the I-124 dosimetry, and the second group will have the I-124 dosimetry performed first followed by the I-131 dosimetry.

The risk of this study is considered very low, and the potential benefits to the patient are considered very high.

DETAILED DESCRIPTION:
Radiopharmacokinetics and Dosimetric Calculations

A tracer dosage of either I-131 or I-124 is first administered to the patient, and the clearance is then followed for the specified period. In the classical approach, the blood is considered the critical organ which is irradiated either from the

* particles emitted from activity in the blood itself, or from the
* emissions originating from activity dispersed throughout the remainder of the body. Therefore only two compartments need to be monitored for radioactivity: (a) blood and (b) the whole body. Based on a classical dosimetry approach, the radiation dose to the whole blood in cGy (rads) per MBq I-131 is calculated.

The calculation of the area under these two curves is based on a mathematical fit to the data points using a multiple exponential function. Since the data collection is terminated after 4 days these curves must then be extrapolated to infinity. A very conservative estimate is employed by assuming that the clearance following the final measured data point is based simply on the physical decay. This ignores any biological clearance and results in an overestimation of the area of these tails and hence in the radiation dose per millicurie administered.

Each patient will have the following calculated.

i. Whole body radiopharmacokinetics

ii. Blood radiopharmacokinetics

iii. Whole blood dosimetry

iv. Lesion Kinetics

i. Whole body radiopharmacokinetics

As an alternative to using an external probe to measure the whole body retention, a dual detector gamma camera system can be used. In this case the patient is scanned in the whole body mode in a reproducible geometry while lying supine on the imaging table. This method has been generally accepted for patient-specific whole body dosimetry of I-131 radiolabeled antibodies . Furthermore, it has been shown to yield comparable results with the external probe data . This technique has the following features:

* Simultaneous anterior and posterior images using a high-energy collimator.
* Table height, detector radii, scan length, scan speed, and energy window are standardized and reproduced for each data point.
* Scan speed can be relatively rapid (typically we have used 30 cm/min) so that the data acquisition is completed in approximately 8 minutes.
* Additional scans are performed each day for (1) background, and (2) a counting standard (vial containing about 37 MBq (1 mCi) of I-131).
* Total counts in the image or fixed regions of interest encompassing the entire body are used for the calculation of whole body retention.

Although the images are not used for diagnostic purposes, this approach has the additional advantage that if for some reason there is delayed absorption of the tracer dosage in the stomach, and then the measurement could be repeated at 4 hours.

During the initial 2-hour period following the I-131 administration the patient is not allowed to urinate or defecate. Under these circumstances essentially 100 percent of the dosage will be contained within the patient at these observation points. The initial image is then defined to represent the 100 percent value and subsequent daily measurements are normalized to this value using the formula:

When used in this way, the standard will correct for variations in detector sensitivity from measurement to measurement, as well as for physical decay. Absolute calibrations are not necessary since the patient is used as his/her reference.

The whole body I-124 images will be obtained at the same time points using the PET system. In this case emission imaging will be obtained for 1-2 minutes/bed position for a sufficient number of positions to cover the patient from head to foot. Transmission imaging will also be performed to correct the emission data for attenuation.

ii. Blood pharmacokinetics

The blood samples (3-4 ml in purple top tubes) are counted using scintillation well-detector system. Since we need to determine the activity in these samples, it is necessary to make up a calibration standard, which can be counted at the same time. This involves the addition of a carefully assayed quantity of I-131 (approximately 3.7 MBq - 7.4 MBq {100-200 uCi}) to a total volume of 1000 ml. Such a small concentration is necessary in order to avoid saturating the detector. An alternative that we have implemented in the dosimetry program here at the Washington Hospital Center uses a Ba-133 rod source instead that has been cross-calibrated against the I-131 standard. With its relatively long half-life (10.3 years) and similar gamma emissions, Ba-133 is a suitable replacement for the prepared I-131 standard. At the conclusion of the data acquisition, two 1-ml aliquots of whole blood, and the "standard" are counted. Using this information, it is possible to calculate the % of administered dosage/liter of whole blood at each of the timed samples. A zero time point is calculated by dividing the total dosage by the patient's total blood volume. However, a patient-specific blood volume is not determined, but is assumed to equal 20% of the body weight.

iii. Whole blood dosimetry

The Maximum Treatment Activity (MTA) is then calculated as the activity of I-131, which would deliver a combined beta and gamma dose to the blood component of 200 cGy (200 rads).

This calculation will be performed using the whole body and blood clearance data from both the I-131 and the I-124 biokinetic clearance data. The I-124 data will first be corrected for the difference in half-lives of these two radionuclides so as to generate the "equivalent" I-131 values.

iv. Lesion Kinetics

For those patients in which focal lesion(s) can be visualized the clearance curves and half-lives will be determined from the images for both the I-131 and the I-124 studies. A manually drawn region-of interest (ROI) will be placed around each lesion as visualized on the diagnostic whole body scan performed at 48hrs post administration of the radioiodine. This ROI will then be positioned over the comparable area on each of the scans. A background ROI adjacent to the lesion will also be drawn. The total counts in the lesion after background correction will be determined for each time point. In the case of the PET scans first each PET study will be co-registered to the diagnostic scan using the Hermes image registration tool. The coronal slices will then be added to generate a whole body scan that is "equivalent" to that of I-131. Regions of interest will be defined in the same manner as discussed above. A least squares single exponential fit will be applied to each of the lesion clearance curves. The half-life of the exponential will then be computed and the values derived for I-131 compared with I-124 for each identified lesion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Well-differentiated thyroid carcinoma
* Referred for I-131 dosimetry
* Preparation with Recombinant Human TSH (rh TSH)

Exclusion Criteria:

* < 18 years of age
* Pregnancy or breast feeding
* Inability to comply with instructions
* Simultaneous participation or participation in any other research study within the last month
* A body weight greater than 350 lbs
* A creatinine > 1.5 mg/ml for males and 1.4 mg/ml for females
* Preparation with thyroid hormone withdrawal(THW)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Compare the measurement of radioiodine uptake and clearance in suspected metastatic foci of well-differentiated thyroid cancer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Van Nostrand, MD, Principal Investigator — Director, Nuclear Medicine
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No